CLINICAL TRIAL: NCT01962038
Title: A Combined Training Program for Veterans With Amnestic Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, J. Kaci Fairchild, PhD, Clinical Psychologist, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAI0002AGG
Record Dates: First submitted 2013-08-26; First posted 2013-10-14 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Amnestic Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Aging
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Muscle Stretching Exercises; Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined Aerobic and Resistance Exercise/Cognitive Training (Active Comparator)
  Interventions: Behavioral: Combined Aerobic and Resistance Exercise; Behavioral: Cognitive Training
- Stretching Exercises/Cognitive Training (Active Comparator)
  Interventions: Behavioral: Stretching Exercises; Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: Combined Aerobic and Resistance Exercise — Gym and home based aerobic and resistance exercises
  Arms: Combined Aerobic and Resistance Exercise/Cognitive Training
Behavioral: Stretching Exercises — Gym and home based stretching exercises
  Arms: Stretching Exercises/Cognitive Training
Behavioral: Cognitive Training — Group-based cognitive training

SUMMARY:
The purpose of this study is examine the efficacy of a combination physical exercise and cognitive training program on improving memory in older Veterans with amnestic Mild Cognitive Impairment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of amnestic Mild Cognitive Impairment
* available informant
* visual and auditory acuity to allow neuropsychological testing
* willingness to participate in exercise training + cognitive training for 8 months
* approval of primary provider to participate in exercise trial

Exclusion Criteria:

* current severe psychiatric disorder
* diagnosis of dementia
* history of neurological or system illness affecting CNS function
* acute illness or unstable chronic illness
* current severe cardiac disease
* inability to exercise consistently because of orthopedic or musculoskeletal problems
* morbid obesity
* inability to read, verbalize understanding and voluntarily sign the informed consent

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-05; Primary Completion 2017-07 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 28 weeks in delayed recall of a word list | Baseline, 24 weeks, 28 weeks
Change from Baseline to 28 weeks in Delayed Recall of Names-Face Task | Baseline, 24 weeks, 28 weeks

SECONDARY OUTCOMES:
Non-Cognitive Outcomes (Depression, Sleep, Quality of Life) | Baseline, Time 2, Time 3

OTHER OUTCOMES:
Exercise Assessment | Baseline, Time 2, and Time 3

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K Fairchild, PhD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Derived] Fairchild JK, Myers J, Louras P, Jo B, McNerney MW, Hallmayer J, Yesavage J. Multimodal Exercise and Cognitive Training Program Improves Cognitive Function in Amnestic Mild Cognitive Impairment. Am J Geriatr Psychiatry. 2024 Apr;32(4):463-474. doi: 10.1016/j.jagp.2023.12.002. Epub 2023 Dec 11. PMID 38220592